CLINICAL TRIAL: NCT02855892
Title: A Randomized, Placebo-controlled, Single-blind, Parallel Design, Multi-center, Phase II Clinical Trial to Evaluate the Efficacy and Safety of GV1001 in Patients With Benign Prostatic Hyperplasia (BPH)
Brief Title: A Phase II Clinical Trial to Evaluate the Efficacy and Safety of GV1001 in Patients With BPH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GemVax & Kael (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KG 3/2014
Record Dates: First submitted 2016-08-01; First posted 2016-08-04 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: GV1001; BPH; Benign prostatic hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Saline Solution; GV1001 peptide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (Placebo Comparator): - Placebo, two-week interval, intradermal administration
  Interventions: Other: Placebo
- Study Group 1 (Experimental): - GV1001 0.4 mg, two-week interval, intradermal administration
  Interventions: Drug: GV1001
- Study Group 2 (Experimental): - GV1001 0.56 mg, two-week interval, intradermal administration
  Interventions: Drug: GV1001
- Study Group 3 (Experimental): - GV1001 0.56 mg, four-week interval, intradermal administration
  : Should be visited every two weeks (GV1001 0.56 mg or placebo is administered alternately at every visit.)
  Interventions: Other: Placebo; Drug: GV1001

INTERVENTIONS:
Other: Placebo
  Other Names: Normal Saline 0.9 %
  Arms: Control Group; Study Group 3
Drug: GV1001
  Other Names: Tertomotide
  Arms: Study Group 1; Study Group 2; Study Group 3

SUMMARY:
This clinical trial is designed as a randomized, placebo-controlled, single-blind, parallel design, multi-center, phase 2 clinical trial to evaluate the efficacy and safety of GV1001 in patients with benign prostatic hyperplasia. Eligible subjects are randomized into a group out of the three study groups and a placebo group after four weeks of placebo run-in period. Placebo run-in period is concurrently proceeded as a wash-out period for previous treatment of benign prostatic hyperplasia, and a placebo is administered intradermally twice with two-week interval during this period. After that, the randomized subjects receive a study drug and a placebo intradermally seven times with two-week interval by visiting at Week 0, 2, 4, 6, 8, 10, and 12. After the treatment period, the subjects additionally visit at Week 13 and 16, and the efficacy is evaluated at Week 4, 8, 12, 13, and 16, and the safety is evaluated over the 16-week period.

DETAILED DESCRIPTION:
Patients will be randomized equally between the four arms.

1. Control group (placebo, two-week interval): 38 subjects
2. Study group 1 (GV1001 0.4 mg, intradermal administration, two-week interval): 38 subjects
3. Study group 2 (GV1001 0.56 mg, intradermal administration, two-week interval): 38 subjects
4. Study group 3 (GV1001 0.56 mg, intradermal administration, four-week interval): 38 subjects

ELIGIBILITY:
[Inclusion Criteria]

All of the following criteria should be satisfied to be enrolled in this clinical trial.

1. A male at 50 years of age and older
2. A patient who satisfies the following clinical signs and symptoms of benign prostatic hyperplasia

   ① A patient with a volume of prostate gland (TRUS) > 30 cc

   ② A patient with moderate to severe lower urinary tract symptoms with IPSS ≥ 13

   ③ A patient with 5-15 mL/sec of maximum flow rate (Qmax) measured when urine volume was at least 125 mL
3. A patient with PSA level < 10 ng/mL (however, if 4 ng/mL < PSA < 10 ng/mL, a person with a biopsy result, confirming that he does not have prostate cancer)
4. A patient with residual urine volume ≤ 200 mL
5. A patient with intention of not using drugs which may affect benign prostatic hyperplasia (5-alpha reductase inhibitors, drugs similar to LHRH, alpha blockers, alpha-beta blockers, anticholinergics, antidiuretic hormones, diuretics, PDE-5 inhibitors, beta-3 adrenoceptor antagonists, etc.), drugs affecting immune system (steroids, immunosuppressants), or health functional foods which may affect a prostate gland (saw palmetto, etc.) during the clinical trial period
6. A patient has to consent not to participate in other clinical trials as a subject during this clinical trial period.
7. Before enrollment to the study, a patient has to consent to avoid pregnancy by using condoms for 90 days after the end of study participation period and treatment. (However, this is not applied if the patient had vasectomy.) Also, a partner of the patient has to consent to avoid pregnancy by using contraceptive devices or oral contraceptives during the patient's participation in clinical trial and for 90 days after the end of treatment, except if the partner reaches menopause or is surgically sterilized. (Consent should be obtained before visit 4, when necessary.)

[Exclusion Criteria]

If any one of the following is applied, a patient cannot be enrolled in this clinical trial.

1. A patient who has hypersensitivity reactions to ingredients of this drug.
2. A patient who received 5-alpha reductase inhibitors other than a drug used in this clinical trial before randomization (within six months)
3. A patient who received drugs similar to LHRH other than a drug used in this clinical trial
4. A patient who has received an unapproved study drug in the past or the study drug for this clinical trial (One exception: a patient can be enrolled when the drug is considered by an investigator not to affect prostate and urinary function, and the patient is not participating in other ongoing clinical trial.)
5. If diagnosed with prostate cancer in the past or at present
6. A patient who was considered by an investigator to have an influence to an evaluation on urine flow symptoms due to other previous or current diseases besides benign prostatic hyperplasia (e.g., neurogenic bladder, bladder neck contracture, urethral stricture, bladder cancer, malignant tumor in lower urinary tract, etc.)
7. A patient who had surgeries or radiation therapies for prostate gland, bladder or pelvis, or who had invasive treatments for benign prostatic hyperplasia
8. A patient who has severe medical condition which may be cause problem to conduct the clinical trial (e.g., chronic heart failure (CHF), difficult-to-control diabetes (HbA1c > 7%), mental disorder, drug, or alcohol abuse, etc.)
9. A patient with moderate to severe liver hypofunction and severe kidney hypofunction (less than 30 mL/min of creatinine clearance)
10. A patient who receives drugs affecting immune system (e.g., immunosuppressives, steroids for systemic action, etc.)
11. Any other patients who are considered to be ineligible for this study by an investigator

[Inclusion Criteria for Randomization]

1. A patient who satisfies the following clinical signs and symptoms of benign prostatic hyperplasia

   ① A patient with a volume of prostate gland (TRUS) > 30 cc *

   ② A patient with moderate to severe lower urinary tract symptoms with IPSS ≥ 13

   ③ A patient with 5-15 mL/sec of maximum flow rate (Qmax) measured when urine volume was at least 125 mL
2. A patient with residual urine volume ≤ 200 mL
3. A partner of the patient has to consent to avoid pregnancy by using contraceptive devices or oral contraceptives during the patient's participation in clinical trial and for 90 days after the end of treatment, except if the partner reaches menopause or is surgically sterilized.

(* In case that additional TRUS examination has been performed after screening, a decision should be made based on the latest result.)

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of doses of GV1001 by comparing the level of change in IPSS scores in three study groups to a control group. | at Week 0, 4, 8, 12, 13, and 16
  IPSS questionnaire: 7-item questionnaire that measures urinary symptoms, but with an additional, independent eighth question on quality of life. It measures the level of urinary symptoms (including incomplete emptying, frequency, intermittency, urgency, weak stream, straining, and nocturia) reported as the total IPSS score. The first 7 items has a 6-point response scale (0=none/never to 5=almost always/5 or more times) with a total score that can range from 0-35: mild (0-7), moderate (8-19), or severe (20-35). The last item assesses quality of life reported as a Quality of Life assessment index.

SECONDARY OUTCOMES:
Change in volume of prostate gland (TRUS) compared to the baseline | at screening and Week 16
  The amount of change from Transrectal Ultrasonography(TRUS) compared to the baseline
Change in maximum flow rate (Qmax) compared to the baseline | at Week 0, 4, 8, 12, 13, and 16
  The amount of change from Maximum(peak) Urinary Flow Rate compared to the baseline
Change in International Index of Erectile Function (IIEF) compared to the baseline | at Week 0, 4, 8, 12, 13, and 16
  IIEF questionnaire: 15-item, 5 domain scale collected by subject interview, relating to the subjects' experience of erectile function (and other sexual parameters) over the previous 4 weeks.
Change in prostate-specific antigen (PSA) compared to the baseline | at Week 0, 13, and 16
  The amount of change from Prostate-specific Antigen (PSA) compared to the baseline
Change in residual urine volume compared to the baseline | at Week 0, 4, 8, 12, 13, and 16
  The amount of change from Residual Urine Volume compared to the baseline
Change in hormones (testosterone, DHT) compared to the baseline | at Week 0, 4, 8, 12, 13, and 16
  The amount of change from Hormones (Testosterone, DHT) compared to the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Seop Lee, Study Chair — Department of Urology, Dongguk University Gyeongju Hospital
Locations (8):
- South Korea (8):
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Dongguk University Gyeongju Hospital, Gyeongju, Gyeongsangbuk-do
  - Inje University Busan Paik Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Chung-ang University Hospital, Seoul
  - Eulji General Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No